CLINICAL TRIAL: NCT05426057
Title: Scaling a Parenting Evidence Based Intervention (EBI) for Latinx Youth Mental Health in Primary Care
Brief Title: Mental Health in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Guillermo Prado, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20210286; 1R01MH124718-01A1 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Depression, Anxiety; Suicide; Drug Use
Keywords: effectiveness-implementation type 1 hybrid trial; Latinx mental health in primary care; Latinx adolescent; eHealth intervention; Familias Unidas; intervention sustainment; parent-centered; family functioning; sexual risk behavior
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Familias Unidas (Experimental): Participants in this group will receive eHealth Familias Unidas-Mental Health. The intervention consists of nine video parent group sessions, one video adolescent session, and four family sessions (parents participate in a total of 13 sessions, adolescents participate in a total of five sessions) that will be delivered by a facilitator to the parent-child dyad via web-conferencing software across 13 weeks.
  Interventions: Behavioral: eHealth Familias Unidas Mental Health
- Prevention as Usual Control (No Intervention): In this condition, participants will not receive an intervention, only the standard of care services which may include information and referral.

INTERVENTIONS:
Behavioral: eHealth Familias Unidas Mental Health — eHealth Familias Unidas is a program designed to target mental health and suicide ideation and behavior. It focuses on promoting mental health by strengthening family and interpersonal protective factors. The program is provided online over a total of 13 sessions: 9 video parent group sessions, each lasting 20-40 minutes in Spanish and 4 web family sessions lasting 45 minutes in either Spanish or English, depending on participant language preference. The video parent group sessions consist of: 1) culturally syntonic telenovela/soap opera series, 2) videotaped parent group discussions, 3) interactive exercises. Web family sessions will be conducted by a trained pediatric staff member.
  Arms: eHealth Familias Unidas

SUMMARY:
The goal of this study is to evaluate in an effectiveness-implementation type I hybrid trial, an enhanced version of eHealth Familias Unidas for reducing depressive, anxious symptoms and suicide behavior in Hispanic youth. The study will use a randomized rollout design with 18 pediatric primary care clinics in the South Florida area.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male adolescents, who self-identify as Hispanic (or Latino(a))
2. Adolescent between the ages of 12 - 16 years
3. Adolescent living with an adult primary caregiver who is willing to participate
4. Families must have broadband internet access on a device, including (but not limited to) a smartphone, iPad, tablet, computer at their home or other location (e.g., school, library, etc.)
5. Families screening positive on poor family communication (a score of less than 75 on the communication measure; see measures) or youth reporting elevated depressive or anxiety symptom scores (defined as 70 to 90 on the K-CAT) or a history of suicide behavior (ideation or attempts).

Exclusion Criteria:

* Families reporting plans to move out of the South Florida area during the study period.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 468 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in depression symptom severity will be measured using the Kiddie Computerized Adaptive Test (K-CAT®). K-CAT® measures severity on a scale of 0 to 100 with higher scores indicating greater depression symptom severity.
Anxiety symptoms | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in anxiety symptom severity will be measured using the Kiddie Computerized Adaptive Test (K-CAT®). K-CAT® measures severity on a scale of 0 to 100 with higher scores indicating greater anxiety symptom severity.
Suicidality | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in suicidality severity will be measured using the Kiddie Computerized Adaptive Test (K-CAT®). K-CAT® measures severity on a scale of 0 to 100 with higher scores indicating greater suicidality symptom severity.
Change in drug use | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in drug use will be reported as the number of days drug use was reported over the last 90 days.
Center for Epidemiologic Studies Depression Scale (CESD) | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in depression symptoms will be assessed with the CESD. Scores range from 0 to 60 with higher scores indicating the presence of more symptoms.

SECONDARY OUTCOMES:
Change in Family Functioning as assessed by the Parenting Practices Questionnaire | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in family functioning will be reported using nine items from the Parenting Practices Questionnaire . Response range varies based on questions, but most response items range from 0 to 4 with higher values indicating better parenting. Scores range from 0 to 36.
Change in Family Functioning as assessed by the Parent Relationship with Peer Group | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in family functioning will be reported using the Parent Relationship with Peer Group. The Parent Relationship with Peer Group is a six item measure with response items ranging from 0 to 24. Higher scores indicate better outcomes.
Change in Family Functioning as assessed by the Parent-Adolescent Communication Scale | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in family functioning will be reported using the Parent-Adolescent Communication Scale. The Parent-Adolescent Communication Scale is a twenty-item questionnaire with a total score ranging from 20 to 100 with higher scores indicating better communication.
Change in unprotected sexual behavior | Baseline to 3 months, baseline to 6 months, baseline to 18 months
  Change in unprotected sexual behavior will be reported as number of days of sex without a condom as reported over the last 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Prado, PhD, Principal Investigator — University of Miami; C. Hendricks Brown, PhD, Principal Investigator — Northwestern University
Locations (17):
- United States (17):
  - Jessie Trice Community Health Center, Miami, Florida
  - Broward Community Health, Miami, Florida
  - Community Health of South Florida, Miami, Florida
  - Medlife Clinical Research, Miami, Florida
  - Prime Care Health, Miami, Florida
  - Care Resource, Miami, Florida
  - Mailman for Child Devlopment, Miami, Florida
  - Pediatric Mobile Clinic, Miami, Florida
  - UM Pediatric Mobile Clinic, Miami, Florida
  - UM UHealth Pediatrics at the Professional Arts Center, Miami, Florida
  - Borinquean Medical Centers, Miami, Florida
  - Belkys Bravo Clinic, Miami, Florida
  - Nicklaus Children Hospital, Miami, Florida
  - South Florida Pediatric Partners, Miami, Florida
  - Pediatric Consultants of Kendall, P.A., Miami, Florida
  - UHealth Pediatrics at Kendall, Miami, Florida
  - Banyan Health Systems, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estrada Y, Lozano A, Boga D, Tapia MI, Perrino T, Velazquez MR, Forster L, Torres N, Morales CV, Gwynn L, Beardslee WR, Brown CH, Prado G. eHealth Familias Unidas Mental Health: Protocol for an effectiveness-implementation hybrid Type 1 trial to scale a mental health preventive intervention for Hispanic youth in primary care settings. PLoS One. 2023 Apr 18;18(4):e0283987. doi: 10.1371/journal.pone.0283987. eCollection 2023. PMID 37071612